CLINICAL TRIAL: NCT03518853
Title: Phase I/II Study of Short-course Hypofractionated Once-weekly Radiation Therapy (SHORT) for Localized Prostate Cancer
Brief Title: Short Course Radiotherapy for Localized Prostate Cancer
Acronym: SHORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/TMC/0612; CTRI/2016/02/006671 (Registry Identifier: Clinical Trials Registry of India (CTRI))
Record Dates: First submitted 2016-05-11; First posted 2018-05-08 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Adenocarcinoma of Prostate

STUDY DESIGN:
Intervention Model Description: Phase I/II study of radiotherapy fractionation
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Short-course Radiation Therapy (Experimental): Short-course Hypofractionated Once-weekly Radiation Therapy: 35Gy in 5 fractions delivered once a week.
  Interventions: Radiation: Short-course Hypofractionated Once-weekly Radiation Therapy

INTERVENTIONS:
Radiation: Short-course Hypofractionated Once-weekly Radiation Therapy — Eligible patients will be treated with a radiation regimen of 35 Gy in 5 fractions delivered at one fraction per week at 7 day intervals. The dose of radiotherapy is based on the consensus alpha beta ratio of 1.5.

SUMMARY:
Hypofractionated external beam radiotherapy has been clinically used for localized prostate cancer in view of the low estimated alpha/beta ratio of prostate cancer cells. Moderate fraction sizes of <4Gy per fraction has been investigated in several phase II/III studies and has been found to be well tolerated with comparable biochemical control in comparison with standard fractionated dose-escalated regimens. Fraction sizes of > 4 Gy has also been investigated in single center studies. However, its toxicity and disease control outcomes is less well known. In this Phase I/II single arm study the investigators aim to treat non-metastatic prostate cancer with stageT1-T4N0M0 and Prostate Specific Antigen (PSA) <60 ng/ml to a regimen of 35Gy in 5 fractions delivered once a week with a view to determine acute toxicity, biochemical control with PSA and late toxicity.

DETAILED DESCRIPTION:
There is robust evidence to suggest that prostate cancers are slow growing with long tumor doubling times. Evidence accumulated from reported results of several thousands of patients suggest that unlike epithelial malignancies, the alpha/beta ratio for prostate cancer is low, in the range of 1.5 compared to 10. From the radiobiological standpoint, this means that instead of conventional daily fraction sizes of 1.8-2Gy, prostate cancer will be equally well if not better approached with larger fraction sizes. Based on this derivation several single arm and randomized studies have been started. Some have already been reported. They show quite uniformly that hypofractionated radiotherapy using fraction sizes of 2.6-3.1 Gy/fraction with appropriate modifications in the total dose is safe and effective. Therefore the paradigm of radiotherapy treatment of prostate cancer is shifting from 37-40Fractions delivered over 7-8 weeks to shorter courses delivered in 20-28fractions delivered over 4-5 weeks.

Taking this approach further it has been hypothesized that the schedule may be modified further and the total number of treatments can be reduced to 4-7 fractions delivered in a spaced schedule over 2-5 weeks. There are already 6-7 published reports of non-randomized cohorts treated with such schedules delivered using Image Guided Intensity modulated Radiation Therapy (IG-IMRT) or stereotactic radiotherapy (SBRT) techniques for localized risk cancers. Preliminary results from these studies show excellent safety and efficacy. These results have considerable implications. If the treatment of prostate cancer can be safely and effectively truncated from 37-40 fractions over 8 weeks to only 4-7 treatments delivered over 2-5 weeks, it results in better patient convenience, compliance, cost savings and also a significant sparing of healthcare resources. All of these are of great importance in countries like India.

The short course hypofractionated schedules have so far been mainly tried in selected risk groups, and have not previously been used in India. The investigators intend to perform a phase I/II study to test the safety and efficacy of a schedule of once weekly hypofractionated radiotherapy. The study population will be 30 patients with localized prostate cancer (T1-T4N0M0) with a PSA <60 ng/ml. The patients will receive image-guided radiotherapy (IGRT) delivering 5 fractions of 7Gy at weekly intervals. Androgen deprivation therapy will be done according to standard criteria based on risk stratification. The primary endpoint of this study is the incidence of acute grade 2 or more side-effects. The secondary endpoints will be biochemical control at 3 years and late grade 2 side-effects at 2 years. Side effects will be monitored according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4. Quality of life assessments will be done using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 and PR25 questionnaires at baseline, treatment completion, 3 and 6 months post treatment.

If found safe and effective, this schedule of treatment will lead to phase I studies comparing this schedule with standard fractionation or more moderate hypofractionation schedules.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma.
* History/physical examination with digital rectal examination of the prostate within 8 weeks prior to registration
* Histological evaluation of prostate biopsy with assignment of a Gleason score to the biopsy material.
* Clinical stage T1-T4N0M0 (AJCC 7th edition). Staging demands a multiparametric MRI of the pelvis a CT or MRI of the abdomen for T3/T4 tumors or PSA >10 a whole body bone scan for T3/T4 tumors or PSA >10
* PSA < 60 ng/mL within 180 days prior to registration. PSA should not be obtained for at least 10 days after prostate biopsy.
* WHO performance status 0-1
* Age ≥ 18
* Patient must sign study specific informed consent prior to accrual.

Exclusion Criteria:

* Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy unless continually disease free for a minimum of 5 years.
* Previous radical surgery (prostatectomy) or cryosurgery for prostate cancer
* Previous pelvic irradiation in any form.
* Previous hormonal therapy of more than 180 days duration prior to registration.
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Severe, active comorbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol. (Patients on Coumadin or other blood thinning agents are eligible for this study.)
  * Renal insufficiency with a creatinine clearance of <30ml/min

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-12; Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Acute Gastrointestinal and Genitourinary toxicity as assessed by National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 | Day 29
  To determine the rates of acute gastrointestinal and genitourinary toxicity according to NCI CTCAE v4.0.

SECONDARY OUTCOMES:
Biochemical control (with measurement of Prostate Specific Antigen measured in ng/ml) | 3 years
  To determine the incidence of biochemical control (with measurement of prostate specific antigen) at 3 years. Failure is defined by the Phoenix criteria of nadir PA value in ng/ml + 2 ng/ml.
Incidence of Late Gastrointestinal Toxicity as assessed by NCI CTCAE v4.0 | 3 years
  the incidence of late gastrointestinal toxicity according to NCI CTCAE v4.0 as assessed at 3 years.
Incidence of Late Genitourinary Toxicity as assessed by NCI CTCAE v4.0 | 3 years
  To determine the incidence of late genitourinary toxicity according to NCI CTCAE v4.0 as assessed at 3 years.
Assessing the Quality of Life by measuring patient reported outcomes using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 questionnaire | 3 years
  To evaluate the quality of life using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30 questionnaire and measure the impact of this regimen of radiotherapy on the global health status, functional scales and all general symptom scores on a scale of 0 to 100 (higher score in global and functional scales representing better quality-of-life, while higher sores on symptom scales representing more symptoms). A scale difference of 10 or more would be considered clinically meaningful in any domain.
Assessing the Quality of Life by measuring patient reported outcomes using European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) PR25 questionnaire | 3 years
  To evaluate the quality of life using the PR25 questionnaire and measure the impact of this regimen of radiotherapy on the prostate cancer related urinary, bowel and hormonal therapy related scores on a scale of 0 to 100 (higher score on symptom scales representing more symptoms). A scale difference of 10 or more would be considered clinically meaningful in any domain.

CONTACTS AND LOCATIONS:
Overall Officials: Indranil Mallick, MD, Principal Investigator — Tata Medical Center
Locations (1):
- Tata Medical Centre, Kolkata, WestBengal, India

IPD SHARING:
Plan to Share IPD: Undecided
Once appropriate authorities approach and once clearance of local authorities is received, data could be shared